CLINICAL TRIAL: NCT06448858
Title: Effect of Body Composition on Some Blood Minerals Status in Obese and Overweight Adolescent; Cross Sectional Study
Brief Title: Minerals Status in Relation to Overweight and Obese Adolescent
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Hussien Abdelmoneim Hassan, Resident doctor, Assiut University
Other Study IDs: Minerals in Adolescent
Record Dates: First submitted 2024-05-16; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Mineral Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese: Patients with BMI more than 30
  Interventions: Diagnostic Test: serum Mn, Se, iron, Cu & Zn levels
- Overweight: Patients with BMI 25-30
  Interventions: Diagnostic Test: serum Mn, Se, iron, Cu & Zn levels
- Control: Patients with BMI less than 25
  Interventions: Diagnostic Test: serum Mn, Se, iron, Cu & Zn levels

INTERVENTIONS:
Diagnostic Test: serum Mn, Se, iron, Cu & Zn levels — Evaluate the concentration of serum Mn, Se, iron, Cu & Zn levels in obese and overweight adolescents.

SUMMARY:
Evaluation of the concentration of serum Mn, Se, iron, Cu & Zn levels in obese and overweight adolescents, Correlate the body composition parameters with these minerals' concentration, Study the association between the metabolic risk factors and the disturbance in minerals levels in these patients.

DETAILED DESCRIPTION:
Obesity in the population tends to be a notable public health threat on the global scale . individuals with higher body mass index (BMI) are considered to have a lower life expectancy . Among the obesity-related indicators, visceral adipose tissue (VAT) is acknowledged an emerging and sensitive predictor for the risk of metabolic syndrome and cardiovascular disease . Therefore, adverse VAT accumulation can influence metabolic health in the population, and its related risk factors should be further investigated.

Micronutrients in obese people are explored because of an excess energy consumption, and therefore, an inadequate intake of trace elements and minerals. This imbalance among energy consumption and the intake is known as hidden hunger. Obesity can lead to nutritional metabolic disorders, in which the general state of trace elements and minerals are altered.

Only a few studies on child and adolescents obesity concerned Trace Elements (TE). TE is involved in the pathogenesis of obesity and obesity related diseases. We tried to assess trace elements status [ Manganese (Mn), selenium (Se) copper (Cu),zinc (Zn)] in obese children and their relationships with VAT and metabolic risk factors of obesity.

Manganese (Mn) is an essential trace element . It plays an important role in fat metabolism.

Selenium (Se) is an essential micronutrient that acts as an antioxidant and possesses multiple metabolic properties.

Copper (Cu) is a trace element that is vital. Cu has been reported to play a role in fat metabolism.

Zinc (Zn) plays an important role. Its deficiency impairs growth, metabolism and immunity.

Iron (Fe) is an essential trace element to sustain all forms of life. Existing research indicates iron deficiency is one of the comorbidities associated with obesity .

ELIGIBILITY:
Inclusion Criteria:

1. Patients in adolescent age (12-18 years old)
2. Patients with BMI over 25.

Exclusion Criteria:

1. Patients younger than 12 years old or older than 18 years old.
2. Patients with history of chronic use of mineral and /or vitamin supplements .
3. Patients with syndromal obesity , endocrine disorder and history of any chronic diseases ,
4. Patients under special diets or chronic use of medication .

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Normal,overweight and obese adolescents
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
concentration of serum Manganese | 1 year
  Evaluate the concentration of serum Mn levels in obese and overweight adolescents.
Concentration of serum selenium | 1 year
  Evaluate the concentration of serum Se levels in obese and overweight adolescents.
Concentration of serum Iron | 1 year
  Evaluate the concentration of serum Iron levels in obese and overweight adolescents.
Concentration of serum copper | 1 year
  Evaluate the concentration of serum Cu levels in obese and overweight adolescents.
Concentration of serum Zinc | 1 year
  Evaluate the concentration of serum Zn levels in obese and overweight adolescents.

SECONDARY OUTCOMES:
BMI and its relation to mineral levels | 1 year
  Correlate the BMI with these minerals' concentration.
Visceral fat and it's relation to mineral levels | 1 year
  Correlate Visceral fat with these minerals' concentration.
Basal metabolic rate and it's relation to mineral levels | 1 year
  Correlate basal metabolic rate with these minerals' concentration.
Body fat percentage and it's relation to mineral level | 1 year
  Correlate body fat percentage with these minerals' concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Bluher M. Obesity: Global epidemiology and pathogenesis. Nat. Rev. Endocrinol. 2019;15:288-298. doi: 10.1038/s41574-019-0176-8. [PubMed] [CrossRef] [Google Scholar] — https://www.nature.com/articles/s41574-019-0176-8
- See also: Liu B., Du Y., Wu Y., Snetselaar L.G., Wallace R.B., Bao W. Trends in obesity and adiposity measures by race or ethnicity among adults in the United States 2011-18: Population based study. BMJ. 2021;372:n365. doi: 10.1136/bmj.n365. [PMC free article] [ — https://www.bmj.com/content/372/bmj.n365.short
- See also: Li Y., Schoufour J., Wang D.D., Dhana K., Pan A., Liu X., Song M., Liu G., Shin H.J., Sun Q., et al. Healthy lifestyle and life expectancy free of cancer, cardiovascular disease, and type 2 diabetes: Prospective cohort study. BMJ. 2020;368:l6669. doi: — https://www.bmj.com/content/368/bmj.l6669.abstract